CLINICAL TRIAL: NCT00630045
Title: A Phase III Study of Surgery in Combination With Neoadjuvant Chemotherapy of Oxaliplatin Plus Capecitabine in Colorectal Cancer With Respectable Liver Metastasis
Brief Title: Phase 3 Study of Surgery Combined With Neoadjuvant Chemotherapy(XELOX) in Colorectal Cancer With Resectable Liver Metastasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University (Other); Sanofi (Industry)
Responsible Party: Yeying Jiang/Associate professor, Peking University People's Hospital,Department of General Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXALIC
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-02

CONDITIONS: Colorectal Cancer; Resectable Liver Metastasis
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Neoadjuvant Therapy; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 2~3 cycles of neoadjuvant chemotherapy before resection of liver metastasis
  Interventions: Drug: neoadjuvant chemotherapy with oxaliplatin and capecitabine; Procedure: resection of liver metastasis
- 2 (Active Comparator): no neoadjuvant chemotherapy, resect the liver metastasis directly
  Interventions: Procedure: resection of liver metastasis

INTERVENTIONS:
Drug: neoadjuvant chemotherapy with oxaliplatin and capecitabine — oxaliplatin: 130mg/m2, d1(Q3w) capecitabine:1000mg/m2 bid, d1-14(Q3w)
  Arms: 1
Procedure: resection of liver metastasis — surgery with the aim of R0 resection

SUMMARY:
This study aims to discuss the efficacy and safety of neoadjuvant chemotherapy with XELOX regimen (oxaliplatin plus capecitabine) .

DETAILED DESCRIPTION:
Liver metastasis is the most important prognostic factor of colorectal cancer. Reasonable multidisciplinary therapy might improve the prognosis of patients with liver metastasis. Surgery has been the first choice under such situation. Recently, neoadjuvant chemotherapy has also shown its value in unresectable liver metastasis, for it can increase the chance of R0 resection and give some clues to chemosensitivity of agents. However, for those resectable lesions, the role and safety of neoadjuvant chemotherapy has yet to be confirmed. so we design this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal cancer with liver metastasis(all patients should have the pathological report of colorectal cancer. The chances of hepatocellular carcinoma or metastasis from other primary lesions should be excluded. )
2. Liver metastasis should be resected with R0 resection and to save enough normal liver tissue
3. Anticipated liver resection: for normal liver, ﹤70%; for liver with cirrhosis, ﹤50%
4. No metastasis of other organs or lymph nodes in abdominal cavity
5. No previous use of oxaliplatin and capecitabine, or previous adjuvant treatment ended more than 6 months
6. Age 18 to 75 years old
7. Karnofsky performance status ≥70
8. Life expectancy of ≥3 month
9. Bilirubin level < 1.5mg/dL
10. Serum creatinine <1.0 times ULN
11. Absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl
12. Having signed informed consent

Exclusion Criteria:

1. previous use of oxaliplatin or fluorouracil-based chemotherapy in 6 months.
2. No R0 resection or not enough normal liver tissue left
3. previous radiotherapy of target lesions
4. accompanied with unresectable other metastasis or malignant pleural fluids or ascites.
5. complete or uncompleted liver obstruction
6. peripheral neuropathy(NCI-CTC grade 1 or more)
7. mental disturbance neuropathy that influence the cognition, including brain metastasis
8. other serious disease such as uncontrollable active infection, heart infarction with 1 year, un controlled hypertension, arrhythmia with high risk, or unstable heart infarction,heart failure, coronary artery disease, myocardial infarction within the last 6 months
9. Other previous malignancy within 5 year, except non-melanoma skin cancer
10. accompany with other anti-tumor therapies,including immune therapy, intervention or injection with chemotherapeutical agents into serous cavity, or participating other clinical trials.
11. Pregnancy or lactation period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
disease free survival rate | 3 year

SECONDARY OUTCOMES:
R0 resection rate | at the time of pathological report
survival rate and over survival | 5 year
surgery related mortality | peri-operation period
response rate and safety of XELOX as a neoadjuvant regimen | no time frame

CONTACTS AND LOCATIONS:
Overall Officials: Shan Wang, MD, Principal Investigator — Peking University People's Hospital, Department of General Surgery; Lin Shen, MD, Principal Investigator — Peking University, School of Oncology, Department of GI Oncology
Locations (2):
- China (2):
  - Peking University, School of Oncology, Beijing, Beijing Municipality
  - Peking University, People's Hospital, Beijing